CLINICAL TRIAL: NCT05033444
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, First in Human Study of the Safety, Tolerability and Pharmacokinetics of PRV-002 in Healthy Volunteers.
Brief Title: A First in Human Study of the Safety, Tolerability and Pharmacokinetics of PRV-002 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Odyssey Group International, Inc. (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRV-002-AU-01; PRV-002-AUU-01 (Other: Avance)
Record Dates: First submitted 2021-08-12; First posted 2021-09-02 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Traumatic Brain Injury (TBI)
Keywords: Safety; Tolerability; Pharmacokinetics; PRV-002
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Drugs, Investigational

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, single ascending dose, multi-cohort study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized in a 3:1 ratio of PRV-002 and Placebo.
  The following controls will be employed to maintain the double-blind status of the study:
  Nasal Spray containing active drug and placebo will be indistinguishable in appearance
  Randomization list will be provided to the study center pharmacist for dispensing purposes and kept in the pharmacy, accessible to the pharmacist and authorized personnel only
  PK results for the SRC between cohorts will be presented in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PRV-002 (Experimental): PRV-002 active formulation
  Interventions: Drug: PRV-002
- Placebo comparator (Placebo Comparator): Placebo used is hydroxypropyl beta cyclodextrin (HPβCD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRV-002 — SAD portion: Eligible participants will be randomized to receive a single ascending dose of PRV-002 on study Day 1. Dose escalation will be conducted in a total of 3 cohorts. Within each cohort, 6 participants will be randomized to receive a single dose of PRV-002. The starting dose, dose increments and dose range to be evaluated are based on available nonclinical data. PRV-002 dose levels in the range of 0.133 to 0.533 mg/kg (based on a 60kg participant) will be investigated.
  MAD portion: Eligible participants will be randomized to receive a multiple (one dose per day for 5 consecutive days). Dose escalation will be conducted in a total of 2 cohorts. Within each cohort, 6 participants will be randomized to receive of PRV-002. The starting dose, dose increments and dose range to be evaluated are based on available nonclinical data. PRV-002 dose levels in the range of 0.133 to 0.266 mg/kg (based on a 60kg participant) will be investigated.
  Other Names: Experimental drug
  Arms: PRV-002
Drug: Placebo — Placebo used is hydroxypropyl beta cyclodextrin (HPβCD)
  Other Names: Placebo control
  Arms: Placebo comparator

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of different dose levels of PRV-002 in Health Volunteers

DETAILED DESCRIPTION:
This Phase 1 study is designed to assess the safety, tolerabilty and pharmcokinetics of different dose levels of PRV-002 in Healthy Volunteers. The study will evaluate 3 dose levels of the investigational product, PRV-002, in 5 cohorts of 8 healthy volunteers per cohort. In each cohort, 6 volunteers will receive the investigational product and 2 volunteers will receive placebo. Dose levels will be evaluated in a sequential manner starting at the lowest dose level. Cohorts 1 - 3 will receive a single dose of PRV-002 or placebo. Cohorts will receive one dose of PRV-002 or placebo per day for 5 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 55 years of age (inclusive) at screening.
3. Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2, with a body weight (to 1 decimal place) ≥ 50 kg at screening.
4. Be non-smokers (including tobacco, e-cigarettes and marijuana) for at least 3 months prior to first study drug administration.
5. Have a negative test for cotinine at the screening visit and at check-in on Day -1.
6. Medically healthy without clinically significant abnormalities (in the opinion of the Investigator) at the screening visit in the Schedules of

   Assessments (SoA), including:
   1. Physical examination without any clinically significant findings
   2. Systolic BP in the range of 90 to 160 mmHg (inclusive) and diastolic BP in the range of 50 to 95 mmHg (inclusive) after 5 minutes in supine position
   3. Heart rate in the range of 40 to 100 bpm (inclusive) after 5 minutes rest in supine position
   4. Body temperature (tympanic or oral) in the range 35.5°C to 37.7°C (inclusive)
   5. No clinically significant findings in serum chemistry, haematology, coagulation, and urinalysis tests
   6. Triplicate 12-lead ECG (taken after the volunteer has been supine for at least 5 minutes) with a QTcF ≤ 450 msec for males and ≤ 470 msec for females and no clinically significant abnormalities
   7. Pulmonary assessments must be within the normal range (forced expiratory volume in 1 second [FEV1], forced vital capacity [FVC] and FEV1/FVC ratio ≥ 80% of normal values; f forced expiratory flow over the middle one half of the FVC [FEF25-75%] > 75% of predicted)
   8. Oxygen saturation (SpO2) monitor ≥ 95%.
7. Medically healthy without clinically significant abnormalities (in the opinion of the Investigator) at the timepoints indicated in the Schedules of Assessments (SoA), including:

   1. Physical examination without any clinically significant findings
   2. Systolic BP in the range of 90 to 160 mmHg (inclusive) and diastolic BP in the range of 50 to 95 mmHg (inclusive) after 5 minutes in supine position
   3. Heart rate in the range of 40 to 100 bpm (inclusive) after 5 minutes rest in supine position
   4. Body temperature (tympanic or oral) in the range 35.5°C to 37.7°C (inclusive)
   5. No clinically significant findings in serum chemistry, haematology, coagulation, and urinalysis tests
   6. Triplicate 12-lead ECG (taken after the volunteer has been supine for at least 5 minutes) with a QTcF ≤ 450 msec for males and ≤ 470 msec for females and no clinically significant abnormalities
   7. Pulmonary assessments must be within the normal range (forced expiratory volume in 1 second [FEV1], forced vital capacity [FVC] and FEV1/FVC ratio ≥ 80% of normal values; f forced expiratory flow over the middle one half of the FVC [FEF25-75%] > 75% of predicted)
   8. Oxygen saturation (SpO2) monitor ≥ 95%.
8. Female volunteers must:

   1. Be of nonchildbearing potential i.e., surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before screening) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause
   2. Have a follicle-stimulating hormone level >40 IU/L at the screening visit),or
   3. If of childbearing potential, must agree not to donate ova, not to attempt to become pregnant and, if engaging in sexual intercourse with a male partner, must agree to use an acceptable method of contraception from signing the consent form until at least 30 days after the last dose of the study drug.
9. Male volunteers must agree not to donate sperm and, if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use an acceptable method of contraception from signing the consent form until at least 90 days after the last dose of study drug.
10. Have suitable venous access for blood sampling.
11. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

    -

Exclusion Criteria:

1. History or presence of significant cardiovascular disease
2. History or presence of significant pulmonary disease
3. History or presence of significant hepatic disease
4. History or presence of significant renal disease
5. History or presence of significant haematological disease
6. History or presence of significant gastrointestinal disease
7. History or presence of significant disease
8. History or presence of significant endocrine disease
9. History or presence of significant immunologic disease
10. History or presence of significant dermatologic disease
11. History or presence of significant or neurological disease
12. No major surgery within the past 3 months determined by the PI to be clinically significant.
13. Absence of any acute illness.
14. Current infection that requires systemically absorbed antibiotic.
15. Current infection that requires systemically absorbed antifungal.
16. Current infection that requires systemically absorbed antiparasitic.
17. Current infection that requires systemically absorbed antiviral medication.
18. Any history of malignant disease in the last 10 years (excludes surgically resected skin squamous cell or basal cell carcinoma).
19. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia.
20. Use of or plans to use systemic immunosuppressive (e.g., corticosteroids, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (e.g., interferon) during the study or within 3 months prior to the first study drug administration.
21. History of risk factors for torsade de pointes (including a family history of long QT syndrome or sudden cardiac death).
22. Known arrythmia
23. Liver function test results elevated more than 1.5-fold above the ULN for gamma glutamyl transferase, bilirubin (total, conjugated and unconjugated), ALP, AST or ALT. Volunteers with ALP and/or ALT/AST above the limits specified may be included, at the discretion of the Investigator, if the levels are unaccompanied by clinical signs and are determined to be normal variants.
24. Liver function test results elevated more than 1.5-fold above the ULN for gamma glutamyl transferase
25. Liver function test results elevated more than 1.5-fold above the ULN for bilirubin (total)
26. Liver function test results elevated more than 1.5-fold above the ULN for bilirubin (conjugated)
27. Liver function test results elevated more than 1.5-fold above the ULN for ALP. Volunteers with ALP above the limits specified may be included, at the discretion of the Investigator, if the levels are unaccompanied by clinical signs and are determined to be normal variants.
28. Liver function test results elevated more than 1.5-fold above the ULN for AST. Volunteers with AST above the limits specified may be included, at the discretion of the Investigator, if the levels are unaccompanied by clinical signs and are determined to be normal variants.
29. Liver function test results elevated more than 1.5-fold above the ULN for ALT. Volunteers with ALT above the limits specified may be included, at the discretion of the Investigator, if the levels are unaccompanied by clinical signs and are determined to be normal variants.
30. Positive test results for active human immunodeficiency virus (HIV-1 or HIV-2) antibodies at the screening visit.
31. Positive test results for active hepatitis B surface antigen (HBsAg) antibodies at the screening visit.
32. Positive test results for active hepatitis C virus (HCV) antibodies at the screening visit.
33. Presence or having sequelae of known to interfere with the absorption, distribution, metabolism, or excretion of drugs such as gastrointestinal, liver, kidney, or other conditions .
34. Estimated creatinine clearance < 60 mL/min using the Cockcroft-Gault formula or serum creatinine more than 1.5-fold above the ULN.
35. History of substance abuse or alcohol abuse (defined as more than 10 standard drinks per week or regularly consuming more than 4 standard drinks on any one day; where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc./Vol], 100 mL wine [12% Alc./Vol], 30 mL spirit [40% Alc./Vol]) within 12 weeks prior to the screening visit.
36. Positive drugs of abuse at the screening visit.
37. Positive drugs of abuse at check-in (Day -1).
38. Positive alcohol breath test results at the screening visit.
39. Positive alcohol breath test results at check-in (Day -1).
40. Use of any prescription or over-the-counter medication (including herbal products, diet aids, and hormone supplements) within 10 days prior to the first study drug administration, - exceptions include use of contraceptives, occasional use of paracetamol (doses of 500 mg up to every 6 hours or 2 g per day maximum for no more than 3 consecutive days), ibuprofen (doses of 400 mg up to every 6 hours or 1.6 g per day maximum for no more than 3 consecutive days), topical ointments, and vitamins or dietary supplements.
41. Consumption of grapefruit or Seville orange (or products containing grapefruit or Seville orange) within 10 days prior to the first administration of study drug.
42. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the trial.
43. Known hypersensitivity to any of the study drug ingredients.
44. Use of any vaccinations within 14 days prior to the first study drug administration.
45. For women of childbearing potential, a positive serum pregnancy test at the screening visit.
46. For women of childbearing potential, a positive urine pregnancy test (with confirmatory serum pregnancy test) at check-in (Day -1).
47. Females who are breastfeeding or planning to breast feed at any time during the study.
48. Donation of blood or plasma within 30 days prior to first study drug administration.
49. Loss of whole blood of more than 500 mL within 30 days prior to first study drug administration.
50. Receipt of a blood transfusion within 1 year of first study drug administration.
51. Participation in another clinical trial of an investigational drug within 60 days of the first study drug administration.
52. Any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Safety endpoint - Evaluation of the Incidence, severity, and relationship of AEs/SAEs (or ADEs/SADEs) (including withdrawals due to AEs (or ADEs)). | Baseline pre-intervention (Day -28 to Day -2 and Day -1); during intervention and immediately afterwards (Day 1); Day 2; and through Day 5.
  AEs/SAEs (or ADEs/SADEs) to be recorded as written descriptions on case report forms
Safety endpoint - Change from baseline in physical examination findings (Full) | Baseline pre-intervention Day -28 to -2.
  Full physical exam including general appearance, head, ears, eyes, nose and throat, neck (including thyroid and lymph nodes), respiratory system, cardiovascular system, gastrointestinal system, renal system, neurological condition, musculoskeletal system, skin and any other focused assessments suggested by the presence of specific symptoms and measured by written descriptions.
Safety endpoint - Change from baseline in physical examination findings (symptom directed) | Baseline pre-intervention Day -1 and and Day 1; Day 2
  Symptom-directed physical examination (focused assessments suggested by the presence of specific symptoms) will be performed if clinically indicated, as determined by the Investigator. The pre-dose physical examination assessment should be performed on the scheduled day, at any time prior to dosing. All other physical examinations will be performed within ± 1 hour of the nominated timepoint. Measured by written descriptions.
Safety endpoint - Change from baseline in vital signs (including changes from baseline in SpO2). | Baseline pre-intervention between Day -28 to -2; Day 1 pre-intervention; Day 1 at 0.5hr, 1hr, 2hr, 6hr; Day 2 at 24 hr post intervention; Day 5
  SpO2 measured as percent of oxygen (%)
Safety endpoint - Change from baseline in vital signs (including changes from baseline in blood pressure). | Baseline pre-intervention between Day -28 to -2; Day 1 pre-intervention; Day 1 at 0.5hr, 1hr, 2hr, 6hr; Day 2 at 24 hr post intervention; Day 5
  Blood pressure measured for systolic and diastolic pressure as mm of mercury.
Safety endpoint - Change from baseline in vital signs (including changes from baseline in heart rate). | Baseline pre-intervention between Day -28 to -2; Day 1 pre-intervention; Day 1 at 0.5hr, 1hr, 2hr, 6hr; Day 2 at 24 hr post intervention; Day 5
  Heart rate measured as beats per minute (BPM)
Safety endpoint - Change from baseline in vital signs (including changes from baseline in respiration rate). | Baseline pre-intervention between Day -28 to -2; Day 1 pre-intervention; Day 1 at 0.5hr, 1hr, 2hr, 6hr; Day 2 at 24 hr post intervention; Day 5
  Respiration rate measured as breaths per minute
Safety endpoint - Change from baseline in vital signs (including changes from baseline in body temperature). | Baseline pre-intervention between Day -28 to -2; Day 1 pre-intervention; Day 1 at 0.5hr, 1hr, 2hr, 6hr; Day 2 at 24 hr post intervention; Day 5
  Body temperature measured as degrees Celsius (C)
Safety endpoint - Changes from baseline in lung spirometry. | Baseline pre-intervention between Day -28 to -2; Day 1 pre-intervention; Day 1 at 0.25hr, 1hr, 10hr; Day 2 at 24 hr post intervention; Day 5
  Lung spirometry measured as the ratio of forced expiratory value (FEV1)/ forced vital capacity (FVC) and reported as percentage (%)
Safety endpoint - Change from baseline in ECG parameters of heart rate | Baseline pre-intervention; during intervention and immediately afterwards (Day 1); Day 2; and through Day 5.
  Heart ratel measured beats per minute (BPM)
Safety endpoint - Change from baseline in ECG parameters of PR interval, QRS interval, and QT interval | Baseline pre-intervention between Day -28 to -2; Day -1; Day 1 pre-intervention; Day 1 at 0.5hr, 2hr, 6hr; 12hr; Day 2 at 24 hr post intervention; Day 5
  PR interval, QRS interval, and QT interval as measured in milliseconds (ms)
Safety endpoint - Change from baseline in hematocrit values | Baseline pre-intervention between Day -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24 hr post intervention; Day 5
  Hematocrit measured as the percentage of red blood cells in whole blood (%)
Safety endpoint - Change from baseline in hemoglobin values | Baseline pre-intervention between Day -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24 hr post intervention; Day 5
  Hemoglobin measured as the amount of hemoglobin in whole blood measured as grams per deciliter (g/dL)
Safety endpoint - Change from baseline in Red Blood Cell (RBC) indices | Baseline pre-intervention between Day -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24 hr post intervention; Day 5
  RBC measured as the number of million RBCs per microliter (mcL) of blood
Safety endpoint - Change from baseline in Thrombocyte Count (Platelets); White Blood Cells (WBC); Basophils; Eosinophils; Lymphocytes; Monocytes; and Neutrophils. | Baseline pre-intervention between Day -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24 hr post intervention; Day 5
  Platelets measured as the number of cells per microliter (mcL) of blood
Safety endpoint - Change from baseline in the blood hormone level of Dehydroepiandrosterone-sulfate (DHEAS) | Baseline pre-intervention Day -1; Day 1 at 6hr; Day 2 at 24 hr; Day 5
  Dehydroepiandrosterone sulfate (DHEAS) measured as the number of micrograms per deciliter (µg/dL) of blood
Safety endpoint - Change from baseline in the blood hormone level of dihydrotestosterone (DHT) | Baseline pre-intervention Day -1; Day 1 at 6hr; Day 2 at 24 hr; Day 5
  Dihydrotestosterone (DHT) measured as the number of nano moles per liter (nmol/L) of blood
Safety endpoint - Change from baseline in the blood hormone level of luteinizing hormone (LH) | Baseline pre-intervention Days -28 to -2
  Luteinizing hormone (LH) measured as the number of International units per liter (IU/L)
Safety endpoint - Change from baseline in the blood hormone level of dehydroepiandrosterone sulfate (DHEAS) | Baseline pre-intervention Day -1; Day 1 at 6hr; Day 2 at 24 hr; Day 5
  Dehydroepiandrosterone sulfate (DHEAS) measured as the number of micrograms per deciliter (mcg/dL)
Safety endpoint - Change from baseline in the blood hormone level of thyroid stimulating hormone (TSH) | Baseline pre-intervention Day -1; Day 1 at 6hr; Day 2 at 24 hr; Day 5
  Thyroid stimulating hormone (TSH) measured as the number of milli-international units per liter (mIU/L)
Safety endpoint - For postmenopausal women only, change from baseline in the blood hormone level of follicle-stimulating hormone (FSH) and human chorionic gonadotropin (hGH) | Baseline pre-intervention Day -1; Day 1 at 6hr; Day 2 at 24 hr; Day 5
  Follicle-stimulating hormone (FSH) and human chorionic gonadotropin (hGH) measured as the number of milli-international units per milliliter (mIU/mL)
Safety endpoint - Change from baseline in the blood hormone level of free thyroxine (FT4), testosterone, and dihydrotestosterone (DHT) | Baseline pre-intervention Day -1; Day 1 at 6hr; Day 2 at 24 hr; Day 5
  Free thyroxine (FT4), testosterone, and dihydrotestosterone (DHT) measured as the number of nanograms per deciliter (ng/dL)
Safety endpoint - Change from baseline in the blood hormone level of progesterone | Baseline pre-intervention Day -1; Day 1 at 6hr; Day 2 at 24 hr; Day 5
  Progesterone measured as the number of nanograms per miiliiliter (ng/mL)
Safety endpoint - Change from baseline in the blood hormone level of estradiol (E2) and free trilodothyronine (FT3) | Baseline pre-intervention Day -1; Day 1 at 6hr; Day 2 at 24 hr; Day 5
  Estradiol (E2) and free trilodothyronine (FT3) measured as the number of picograms per milliliter (pg/mL)
Safety endpoint Change in baseline in clotting factors Partial thromboplastin time (aPTT) and Prothrombin time (PT) | Baseline pre-intervention between Day -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24 hr post intervention; Day 5
  Partial thromboplastin time (aPTT) and Prothrombin time (PT) measured as time to clot in seconds (sec)
Safety endpoint - Change from baseline in the clotting factor Fibrinogen | Baseline pre-intervention between Day -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24 hr post intervention; Day 5
  Fibrinogen measured as the number of milligrams per deciliter (mg/dL)
Safety endpoint - Change from baseline in the clotting factor International Normalized Ratio (INR) | Baseline pre-intervention between Day -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24 hr post intervention; Day 5
  International Normalized Ratio (INR) measured as the ratio of patient PT/control PT
Safety endpoint - Change from baseline in urinalysis parameters bilirubin, blood, glucose, nitrites, protein, and urobilinogen | Post dose Day 1 at 0 to 6hr, 6 to 12hr, and 12 to 24hr
  Bilirubin, blood, glucose, nitrites, protein, and urobilinogen measured as the number of milligrams per deciliter (mg/dL)
Safety endpoint - Change from baseline in urinalysis parameter ketones | Post dose Day 1 at 0 to 6hr, 6 to 12hr, and 12 to 24hr
  Ketones measured as the number of millimoles per liter (mmol/L)
Safety endpoint - Change from baseline in urinalysis parameter leukocyte esterase | Post dose Day 1 at 0 to 6hr, 6 to 12hr, and 12 to 24hr
  Leukocyte esterase measured as negative or positive; number of WBCs per high power field
Safety endpoint - Change from baseline in urinalysis parameter pH | Post dose Day 1 at 0 to 6hr, 6 to 12hr, and 12 to 24hr
  pH measured as pH units
Safety endpoint - Change from baseline in urinalysis parameter specific gravity | Post dose Day 1 at 0 to 6hr, 6 to 12hr, and 12 to 24hr
  Specific gravity measured as specific gravity units as a ratio of density of urine/density of water
Safety endpoint - Change from baseline in serum chemistry parameters globulin, protein, and albumin | Baseline pre-intervention Days -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24hr; Day 5.
  Globulin, protein, and albumin measured as grams per deciliter (g/dL)
Safety endpoint - Change from baseline in serum chemistry parameter alkaline phosphatase | Baseline pre-intervention Days -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24hr; Day 5.
  Alkaline phosphatase measured as International units per liter (IU/L)
Safety endpoint - Change from baseline in serum chemistry parameters bicarbonate, chloride, sodium, and magnesium | Baseline pre-intervention Days -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24hr; Day 5.
  Bicarbonate, chloride, sodium, and magnesium measured as milliequivalents per liter (mEq/L)
Safety endpoint - Change from baseline in serum calcium, glucose, phosphate, creatinine, urea, uric acid, bilirubin (conjugated and unconjugated), high density lipoproteins, low density lipoproteins, total bilirubin, total cholesterol | Baseline pre-intervention Days -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24hr; Day 5.
  Calcium, glucose, phosphate, creatinine, urea, uric acid, bilirubin (conjugated and unconjugated), high density lipoproteins, low density lipoproteins, total bilirubin, total cholesterol, triglycerides measured as milligrams per deciliter (mg/dL)
Safety endpoint - Change from baseline in serum chemistry parameters potassium | Baseline pre-intervention Days -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24hr; Day 5.
  Potassium measured as millimoles per liter (mmol/L)
Safety endpoint - Change from baseline in serum chemistry parameters lipase, creatine kinase, lactate dehydrogenase, aspartate aminotransferase, gamma-glutamyl transferase, alanine aminotransferase, and amylase | Baseline pre-intervention Days -28 to -2; Day -1; Day 1 at 6hr; Day 2 at 24hr; Day 5.
  Lipase, creatine kinase, lactate dehydrogenase, aspartate aminotransferase, gamma-glutamyl transferase, alanine aminotransferase, and amylase measured as Units per liter (U/L)
Safety endpoint - Change from baseline in virology parameters HIV-1/-2; HBsAg; HCV; SARS-COV-2 | Baseline pre-intervention Day -28 to -2
  HIV-1/-2; HBsAg; HCV; SARS-COV-2 test results measured as negative or positive
Safety endpoint - Change from baseline in drug screen findings for alcohol | Baseline pre-intervention Day -28 to -2; Day -1
  Alcohol test results measured as percentage (%)
Safety endpoint - Change from baseline in urine drug screen findings for amphetamines, barbiturates, benzodiazepines, cocaine, cotinine, methamphetamines, opiates, phencyclidine, THC, and tricyclic antidepressants | Baseline pre-intervention Day -28 to -2; Day -1
  Urine amphetamines, barbiturates, benzodiazepines, cocaine, cotinine, methamphetamines, opiates, phencyclidine, THC, and tricyclic antidepressants test results measured as nanograms per milliliter (ng/mL)
Safety endpoint - Change from baseline for pregnancy test for serum hCG and urine hCG | Serum pregnancy test Days -28 to -2 and on Day 5; Urine pregnancy test Day -1
  Serum hCG and Urine hCG levels measured in milli-international units per liter (mIU/L)
Safety endpoint - Change from baseline for confirmation of postmenopausal status test for FSH | Baseline pre-intervention on Days -28 to -2
  FSH levels measured in milli-international units per liter (mIU/L)

SECONDARY OUTCOMES:
Plasma pharmacokinetics - Cmax | Samples collected on Day 1 pre-dose and at 0.25, 0.5, 1, 1.5, 2. 3, 4, 6, 10, 12hrs; Day 2 at 24 hr; Day 5.
  Plasma PRV-002 Cmax measured as microgram per mL (mcg/mL)
Plasma pharmacokinetics - Tmax | Samples collected on Day 1 pre-dose and at 0.25, 0.5, 1, 1.5, 2. 3, 4, 6, 10, 12hrs; Day 2 at 24 hr; Day 5.
  Plasma PRV-002 time to Cmax
Plasma pharmacokinetics - area under the curve | Samples collected on Day 1 pre-dose and at 0.25, 0.5, 1, 1.5, 2. 3, 4, 6, 10, 12hrs; Day 2 at 24 hr; Day 5.
  Plasma PRV-002 Area under the concentration-time curve from 0 to time of last quantifiable concentration (AUC0-t) measured as min*kBq/mL
Plasma pharmacokinetics - area under the concentration-time curve | Samples collected on Day 1 pre-dose and at 0.25, 0.5, 1, 1.5, 2. 3, 4, 6, 10, 12hrs; Day 2 at 24 hr; Day 5.
  Plasma PRV-002 area under the concentration-time curve from 0 to infinity (AUC0-inf) measured as mg*h/L
Plasma pharmacokinetics - apparent terminal elimination half-life t1/2) | Samples collected on Day 1 pre-dose and at 0.25, 0.5, 1, 1.5, 2. 3, 4, 6, 10, 12hrs; Day 2 at 24 hr; Day 5.
  Plasma PRV-002 apparent terminal elimination half-life (t1/2) measured in minutes or hours
Plasma pharmacokinetics - terminal elimination rate constant (λz) | Samples collected on Day 1 pre-dose and at 0.25, 0.5, 1, 1.5, 2. 3, 4, 6, 10, 12hrs; Day 2 at 24 hr; Day 5.
  Plasma PRV-002 terminal elimination rate constant (λz) measured as elimination rate measured as constant K or Ke ((λz))
Plasma pharmacokinetics total apparent body clearance | Samples collected on Day 1 pre-dose and at 0.25, 0.5, 1, 1.5, 2. 3, 4, 6, 10, 12hrs; Day 2 at 24 hr; Day 5.
  Plasma PRV-002 total apparent body clearance measured as (CL/F)
Plasma pharmacokinetics - apparent volume of distribution | Samples collected on Day 1 pre-dose and at 0.25, 0.5, 1, 1.5, 2. 3, 4, 6, 10, 12hrs; Day 2 at 24 hr; Day 5.
  Plasma PRV-002 apparent volume of distribution measured as (Vz/F)
Urine pharmacokinetics - cumulative amount of unchanged drug excreted in urine | Baseline pre-intervention on Day -1; Day 1 at 0 to 6hr, 6 to 12hr, and 12 to 24 hr.
  Urine PRV-002 cumulative amount of unchanged drug excreted (Ae) in urine measured in micrograms per milliliter (mcg/mL)
Urine pharmacokinetics - renal clearance | Baseline pre-intervention on Day -1; Day 1 at 0 to 6hr, 6 to 12hr, and 12 to 24 hr.
  Urine PRV-002 renal clearance measured as (CLr)

OTHER OUTCOMES:
Exploratory endpoints - PRV-002 metabolites in plasma | Samples collected on Day 1, 2, and 5
  PRV-002 metabolites in plasma measured as micrograms per milliliter (mcg/mL)
Nasal Spray Attributes Questionnaire | Nasal spray attributes questionare completed on Day 1 at 15 minutes post dose
  Nasal Spray Attributes Questionnaire score, based on a scale of 0 to 6, for each immediate attribute assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Ryan, Dr., Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network Pty Ltd,, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.oragenics.com/